CLINICAL TRIAL: NCT02483819
Title: Changes of the Hemodynamic Profiles on Bio Reactance Technique During TURP in Elderly Patients
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2015-0362
Record Dates: First submitted 2015-06-18; First posted 2015-06-29 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Benign Prostate Hyperplasia
Keywords: Elderly patient; NICOM; TURP
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the change of the hemodynamic profiles on bio reactance technique during TURP in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

1) Twenty (ASA status I ~ III) patients, ages 65 to 80 yr old, who were scheduled for transurethral resection of the prostate under spinal anesthesia

Exclusion Criteria:

1. if there were contraindications for spinal anesthesia including hypersensitivity to any local anaesthetics, bleeding diathesis, infections at the puncture sites, or pre-existing neurological disease.
2. history of coronary artery bypass surgery
3. history of dementia
4. have a difficulty in understanding informed consent or refuse to sign the informed consent
5. patients height under 150 cm

Ages: 65 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: elderly patients undergoing transurethral resection of the prostate under spinal anesthesia
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-07-02 (Actual); Primary Completion 2016-02-27 (Actual); Study Completion 2016-02-27 (Actual)

PRIMARY OUTCOMES:
change of the hemodynamic profiles including cardiac index on NICOM during the TURP in elderly patients | change from baseline 1 min before the anesthesia, 10 min after anesthesia, 10 min after surgery, 20 min after surgery, 30 min after surgery, at the end of the surgery
  (Cardiac output, stroke volume, Stroke volume index, Total peripheral resistance, heart rate, blood pressure)

SECONDARY OUTCOMES:
change of the electrolyte | from expected up to 3 months before surgery for preoperative evaluation to expected up to 3 hours after the end of surgery
change of the hemoglobin | from expected up to 3 months before surgery for preoperative evaluation to expected up to 3 hours after the end of surgery
estimated absorbed irrigation fluid during the surgery | during the surgery
  Fluid absorbed = % decrease in sodium x ECF (0.2 x body weight)
incidence of TURP syndrome | followed for the duration of hospital stay, an expected average of 7 days.